CLINICAL TRIAL: NCT03915288
Title: MODERATE CONTINUOUS TRAINING VERSUS HIIT ON CARDIOMETABOLIC AND PSYCHOSOCIAL VARIABLES IN CANCER STADIUM II.CONTROLLED RANDOMIZED TRIAL
Brief Title: MODERATE CONTINUOUS TRAINING VERSUS HIIT IN CANCER STADIUM II.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tolteca (Other)
Responsible Party: Principal Investigator, Javier Eliecer Pereira Rodriguez, Physiotherapist, specialist in cardiopulmonary rehabilitation, magister in health sciences, university professor., University Tolteca
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: JPereiraRodriguez
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Cancer; Fatigue; Sarcopenia
Keywords: Cancer; Aerobic exercise; High intensity training; Force
MeSH Terms: conditions — Neoplasms; Fatigue; Sarcopenia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 1573 cancer patients, who, after the exclusion criteria, 812 patients with stage II cancer finally started the investigation and were organized into 3 groups. The present, was distributed with a basic probabilistic sampling by means of a table of random numbers, whose order was randomized through the program Microsoft Excel 16.0, being the experimental group 1 with 270 participants (MICT + strength training), 275 participants in experimental group 2 (HIIT + strength training) and control group with 267 (verbal recommendations on exercise, diet, follow-up via telephone call and carrying out activities of daily living).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group continuous training at moderate intensity (Experimental): Training program lasting 36 weeks with assistance 3 times a week with 70 minutes per intervention, where 10 minutes were warm up (breathing exercises, walking, stretching), 30 minutes of continuous aerobic training at moderate intensity - MICT (60 -80% FCM), 20 minutes of strength training (40-60% maximum strength) with dumbbells and theraban. And the last 10 minutes were for cooling (exercises coordination, balance, walking and breathing exercises).
  Regarding the MICT training, this was done with fast walk or jog in endless band with the floor tilted to reach the desired intensity. Also by bicycle, rowing and elliptical. During the entire intervention the participants was monitored by a Polar Multisport RS800CX, oximetry and with the Borg scale to avoid exceeding the training intensity (60-80% FCM, 6 to 8 Borg).
  Interventions: Other: Group continuous training at moderate intensity
- Group high Intensity Interval Training (Experimental): Training program lasting 36 weeks with assistance 3 times a week with 70 minutes per intervention, where 10 minutes were warm up (breathing exercises, walking, stretching), 30 minutes of continuous aerobic training at moderate intensity (60 -80% FCM), 20 minutes of strength training (40-60% maximum strength) with dumbbells and theraban. And the last 10 minutes were for cooling (exercises coordination, balance, walking and breathing exercises).
  Concerning the HIIT training, it consisted of an intensity of interval training. That is, the participants who underwent 30 minutes of aerobic exercise consisted of a protocol created for this experimental group, which we named 30-30. 30 seconds at moderate intensity (60-80% FCM) and 30 seconds at high intensity (80-90%).
  Interventions: Other: Group high Intensity Interval Training
- Group control (Active Comparator): This group did not perform supervised exercise nor were they given exercise recipes or formal intervention programs. Only continued with the usual care and gave directions to maintain a healthy lifestyle based on proper nutrition and usual activities. It is highlighted that in the institutions where the patients of the 3 groups attended, there is not a physical training area supervised by a professional. Therefore, the intervention protocol was not excluded or denied to the participants of the control group, but continuity and supervision was given for investigative purposes to its process and treatment. In addition, none of the 3 groups stopped their medical treatment or that of the other professionals that make up the interdisciplinary team.
  Interventions: Other: Group control

INTERVENTIONS:
Other: Group continuous training at moderate intensity — 70 minutes for intervention, where 10 minutes were warm up (breathing exercises, walking, stretching), 30 minutes of continuous aerobic training at moderate intensity (60-80% FCM), with fast walking or endless tread with the floor inclined to reach the desired intensity. Also on bicycle, rowing and elliptical; Then, 20 minutes of strength training (40-60% maximum strength) with dumbbells and theraban. Ends with 10 minutes of cooling with walking and breathing exercises.
  Arms: Group continuous training at moderate intensity
Other: Group high Intensity Interval Training — 70 minutes for intervention, where 10 minutes were for warm-up (Respiratory exercises, walking, stretching), 30 minutes consisted of an intensity of interval training. That is, the participants who underwent 30 minutes of aerobic exercise consisted of a protocol created for this experimental group that we named 30-30. 30 seconds at moderate intensity (60-80% FCM) and 30 seconds at high intensity (80-90%). ; Then, 20 minutes of strength training (40-60% maximum strength) with dumbbells and theraban. Ends with 10 minutes of cooling with walking and breathing exercises.
  Arms: Group high Intensity Interval Training
Other: Group control — This group did not perform supervised exercise nor were they given exercise recipes or formal intervention programs. Only continued with the usual care and gave directions to maintain a healthy lifestyle based on proper nutrition and usual activities.
  Arms: Group control

SUMMARY:
Introduction: Exercise programs focused on moderate intensity continuous training (MICT) and HIIT (High Intensity Interval Training) are shown as an effective treatment to mitigate the effects of cancer.

Objective: To determine and compare the effects of MICT vs. HIIT on the cardiometabolic and psychosocial variables of the cancer patient.

Methods and materials: Randomized controlled trial of 3 years and 4 months in participants with stage II cancer divided into 3 groups (MICT, HIIT and control group). Risk factors, blood samples for glycemia and lipid profile were identified. In addition, 6-minute walk, stress test for maximum heart rate (HRM), anthropometry, quality of life, fatigue, sarcopenia, depression, anxiety, clinical and hemodynamic parameters. All tests were done before and after 36 training sessions of 70 minutes, 3 times a week.

DETAILED DESCRIPTION:
MATERIALS AND METHODS

This investigation was a randomized clinical trial, which included the participants with stage II cancer who were randomly assigned to the MICT group (Experimental Group 1), HIIT (Experimental Group 2) or group of usual considerations (Control Group). The present, was distributed with a basic probabilistic sampling by means of a table of random numbers, whose order was randomized through the program Microsoft Excel 16.0, being the experimental group 1 with 270 participants (MICT + strength training), 275 participants in experimental group 2 (HIIT + strength training) and control group with 267 (verbal recommendations on exercise, diet, follow-up via telephone call and carrying out activities of daily living). The execution period was 3 years and 4 months (November 2015 - February 2019) to obtain the following attributes:

Characteristics of the participants The participants contained similar characteristics from the point of view of: Cancer stage, ejection fraction, functional class, glucose, lipid profile, muscle percentage, fat and BMI (body mass index), abdominal circumference, overweight, obesity, prevalence of diabetes, hypertension (HBP), cardiovascular risk factors and in some cases surgical intervention. In addition, all participants presented "High risk" according to the stratification proposed by the American Association of Cardiopulmonary Rehabilitation.

Blind methodology A simple blind clinical study was carried out, in which the participants were initially evaluated by a non-investigating professional (oncology doctor of the Oncology service). Subsequently, the participants accessed a database in Microsoft Excel 16.0 exclusively with an identification number that allowed the blinding of the investigators. As they were entering the randomized clinical trial, he/she was randomly located in one of the three groups (MICT-HIIT-GC), according to how the computer generated the group location sequence. All participants and professionals, including researchers, were blinded throughout the protocol.

For groups 1 and 2 (MICT-HIIT), the investigators prepared the questionnaires and tests without them knowing the assignment of each patient. For experimental groups 1 and 2, the evaluating authors were D. P-F. - C. Q-G .; and X. V-B. - K. S-P. respectively.

After the tests, the participants were suggested to approach the main investigator (J. P-R) to inform them of their schedule and the start date of the training program. However, we emphasize that from the initial exams until the end of the training program, the authors did not establish a conversation on the subject with the participants or the therapists. Exclusively, the investigators carried out questionnaires, tests and pre and post-training tests and alone, the investigator J. P-R. held regular meetings with the physiotherapists trainers to know and harmonize the training of each group, but not to intimate with the participants or review their data.

After the training program, tests and examinations were performed on the patients of each group to calculate the changes after the training. Taking into account the information gathered before and after, the statistical analyzes for experimental group 1 were carried out by X. V-B. and K. S-P .; for experimental group 2 by D. P-F. and C. Q-G. and for the control group, the investigators J. P-R. and E. G-D. Finally, once the different variables were studied blindly, all the investigators were informed about the groups with their corresponding participants and the results to generate the conclusions all together.

Anthropometric characteristics In all the participants the following data were obtained: Family and personal background using a self-created questionnaire. Also, anthropometric measures (weight, height, body mass index, abdominal circumference, percentage of fat and muscle) using standardized techniques in the Mexican population.

Weight, percentage of fat and muscle were obtained using the digital scale previously calibrated and located on a flat and stable surface, using the indications of the user manual. On the other hand, the height was obtained with a tallimeter placing the participants standing, with the head in the Frankfort plane and the shoulders relaxed to avoid the lordosis and the lower limbs completely against the wall. Having said the above, with these variables the BMI was determined in kg/m-1. Then, with a tape measure and a precision of 1 mm, the measurement of the abdominal circumference was collected.

Clinical and hemodynamic parameters After all the above procedures, blood glucose levels were determined on the first and last day of your training session. The blood sample was taken between 7:00 and 8:00 a.m., after 8-10 hours of fasting. This same sample served to define the levels of cholesterol, triglycerides, low density lipoproteins (LDL) and high density lipoproteins (HDL). In addition, each patient underwent a 2-D (two-dimensional) echocardiography before and after the training program, to visualize the structures, left ventricular ejection fraction (LVEF) and analyze their mobility in real time. In this same evaluation, the functional class of each patient was identified according to the NYHA classification (New York Heart Assosiation); which designates 4 classes (I, II, III and IV) based on the limitations of the participant's physical activity, caused by cardiac symptoms. Similarly, perceived dyspnea and exertion were assessed using the modified Borg scale. The heart rate was detected by the Polar Multisport RS800CX system and the respiratory one, as the systolic and diastolic blood pressure were obtained manually, while the oxygen saturation was obtained with a portable oximeter.

Questionnaires and tests From the beginning, the participants underwent a medical evaluation in the oncology area to understand the participant's current status, sociodemographic, anthropometric and physiological characteristics. On the same day, it was assessed by physiatry and physiotherapy to estimate exercise tolerance through the 6-minute walk test, which was superimposed before and after the 36 training sessions. The protocol for the 6-minute walk test was conducted in accordance with the ATS Statement: Guidelines for the six-minute walk test of the American Thoracic Society.

After this evaluation day, the participants had to return the following day to perform an exercise test according to the Naughton protocol, which is recommended in high-risk patients and whose velocity and inclination in the endless band is by stages 2 minutes. The investigators emphasize that for these tests, the participants was told that he should avoid smoking, drinking drinks or any type of medication that could alter his vital signs or performance during the test.

Ethical considerations The design and development of the research was carried out under the ethical considerations of the Declaration of Helsinki, signature informed consent and under the authorization of the participants, managers, coordinators and ethics committee of the institution.

ELIGIBILITY:
Inclusion Criteria:

* Participants with cancer stadium II
* To sign an informed consent endorsed by the ethics and research committee of the institution.
* Participants with ejection fraction greater than 35%
* Participants do not have any inconvenience when doing the questionnaires, tests and measures that the investigation demands,
* Participants than will can to go 3 times a week for Cardiovascular rehabilitation.

Exclusion Criteria:

* Participants who had severe pain in the lower or upper limbs.
* Unstable angina.
* Heart rate >120 bpm (beats per minute) at rest.
* Systolic blood pressure >190 mmHg.
* Diastolic blood pressure >120 mmHg.
* Participants who had a positive contraindication make exercise were not admitted in the study.
* Participants to show hemodynamic instability without improving during any test or during the intervention process.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1573 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Changes in ejection fraction after 36 training sessions (%) | After 3 month of training (36 training sessions)
  it is the most important measure of cardiac functioning. This value, expressed as a percentage, measures the decrease in the volume of the left ventricle of the heart in systole, with respect to the diastole. The normal values are higher than 45%.
Changes of the maximum heart rate in a effort test after 36 training sessions | After 3 month of training (36 training sessions)
  It is the maximum capacity that the heart has to contract and we determine it by means of an effort test. The Maximum heart rate can be determined by formula or in a effort test (In the present investigation) which consists in mounting the participant in an endless band with an inclination and speed determined according to the protocol for said test. The test is stopped when the participant. indicates that it can not be more or there are electrocardiographic alterations that indicate that it is the participant's maximum.
Changes in the Body weight after 36 training sessions (Kg) | After 3 month of training (36 training sessions)
  How much body weight (kg) pre and post intervention
Changes in the Body Mass Index after 36 training sessions (%) | After 3 month of training (36 training sessions)
  it is a mathematical reason that associates the mass and the size of an individual. it is also known as the Quetelet index. This result is determined by the formula of weight/square size.
Changes in the Abdominal circumference after 36 training sessions (cm) | After 3 month of training (36 training sessions)
  It is the measurement of the distance around the abdomen at a specific point. Abdominal circumference is used to diagnose and monitor abdominal obesity. The values are in centimeters and according to the population to be studied, the measurements must be less than 90cm for men and 80cm for women.
Changes in the Fat percentage after 36 training sessions (%) | After 3 month of training (36 training sessions)
  Percentage of body fat is considered a measure to determine the level of body fat and a high percentage is a risk factor that triggers multiple chronic diseases. This measure can be determined in many ways but in our study it was used by means of bioimpedance. The normal values for men and women depend on the age of the patients and the manufacturer of the scale.
Changes in the Muscle percentage after after 36 training sessions (%) | After 3 month of training (36 training sessions)
  Muscle percentage is considered a measure to determine the level of muscle in the body and a low percentage is a risk factor that indicates sarcopenia and is associated with a decrease in quality of life. This measure can be determined in many ways but in our study it was used by means of bioimpedance. The normal values for men and women depend on the age of the patients and the manufacturer of the scale.
Changes in the levels of Depression and Anxiety after 36 training sessions | After 3 month of training (36 training sessions)
  Psychological alteration that can be determined by the "Hospital Anxiety and Depression Scale". This scale consists of a series of questions for depression and others for anxiety. The final grade is in the range of 1 to 10 and for the diagnosis of depression or anxiety the result must be greater than or equal to 8.
Changes in the levels of force after 36 training sessions | After 3 month of training (36 training sessions)
  Strength is the physical ability to perform a job or a movement. It can be assessed with 1 maximum repetition and the maximum weight the participant manages to lift will be the reference value for his prescription. In addition, muscle strength can be assessed by dynamometry and indicates low, normal or high muscle strength. Their values depend on the age and sex of the participant.
Changes in the levels of Sarcopenia after 36 training sessions | After 3 month of training (36 training sessions)
  Sarcopenia is the degenerative loss of muscle mass and strength as you get older. It is of high prevalence in patients with cancer. Sarcopenia is assessed according to the European Consensus on Sarcopenia (2010) who presented a diagnostic algorithm based on three criteria. Exploration of gait, muscle strength and muscle mass.
  For the first criterion, we use the Short Physical Performance Battery (SPPB). For the second criterion, the muscular strength, the dynamometry test is used (See force section). And in a final criterion, the muscle mass was assessed using the body mass index and the circumference of the calf, taking as a cut-off point the 31 cm.
Changes in the levels of Fatigue after 36 training sessions | After 3 month of training (36 training sessions)
  Fatigue was assessed using the FACT-Fatigue Scale Scale (Fatigue Scale of the Functional Evaluation of Cancer Therapy), which is an inventory of 13 items that assesses the severity of cancer-associated fatigue (FAC) in the last week. with a scale of 0 to 4 and that with higher scores reflect a lower FAC.
Changes in the levels of Quality of life after 36 training sessions | After 3 month of training (36 training sessions)
  For the quality of life, it is necessary to use the questionnaire called EORTC QLQ-C30 (Version 3), which has 30 questions, where each question will go with a score of 1 to 4 and the higher the final result the better the quality of life. participant's life
Changes in the levels of Total cholesterol after 36 training sessions (mg/dl) | After 3 month of training (36 training sessions)
  It is part of the measures to determine the lipid profile of a person and serves to determine different types of dyslipidemia. This item is obtained by means of a blood sample analyzed in a clinical laboratory and the result obtained by a professional for this purpose. Values above 200 mg/dl are indicative of a lipid alteration.
Changes in the levels of Triglycerides after 36 training sessions (mg/dl) | After 3 month of training (36 training sessions)
  It is part of the measures to determine the lipid profile of a person and serves to determine different types of dyslipidemia. This item is obtained by means of a blood sample analyzed in a clinical laboratory and the result obtained by a professional for this purpose. Values above 150 mg/dl are indicative of a lipid alteration.
Changes in the levels of LDL after 36 training sessions (mg/dl) | After 3 month of training (36 training sessions)
  It is part of the measures to determine the lipid profile of a person and serves to determine different types of dyslipidemia. This item is obtained by means of a blood sample analyzed in a clinical laboratory and the result obtained by a professional for this purpose. Values above 100 mg/dl are indicative of a lipid alteration.
Changes in the levels of HDL after 36 training sessions (mg/dl) | After 3 month of training (36 training sessions)
  It is part of the measures to determine the lipid profile of a person and serves to determine different types of dyslipidemia.This item is obtained by means of a blood sample analyzed in a clinical laboratory and the result obtained by a professional for this purpose. Values lower than 40 mg/dl are indicative of a lipid alteration.
Changes in the levels of Glucose after 36 training sessions (mg/dl) | After 3 month of training (36 training sessions)
  It is used to determine blood glucose levels and its high values are indicative for diabetes mellitus. This item is obtained by means of a blood sample analyzed in a clinical laboratory and the result obtained by a professional for this purpose. Values lower than 126 mg/dl are indicative of diabetes mellitus.

SECONDARY OUTCOMES:
Changes in the Estimated maximum oxygen volume after 36 training sessions (ml/kg/min) | After 3 month of training (36 training sessions)
  It is the maximum amount of oxygen that the body can absorb, transport and consume in a given time, is the blood that our body can transport and metabolize. To determine the Vo2 values, the 6-minute walking test is used and to determine the result of the test, formulas are used according to the meters traveled, age, sex, height and weight of the participant. The larger the meters traveled, the greater the vo2.
Changes in the unit of measurement of the metabolic index (METs) after 36 training sessions (ml/kg/min) | After 3 month of training (36 training sessions)
  It is the unit of measurement of the metabolic index (amount of energy consumed by an individual in a resting situation). To determine the METs values, the 6-minute walking test is used and to determine the result of the test, formulas are used according to the meters traveled, age, sex, height and weight of the participant. The larger the meters traveled, the greater the METs.
Changes in the Distance traveled after 36 training sessions (m) | After 3 month of training (36 training sessions)
  Distance traveled in this of 6 minute walk test. The larger the meters traveled, this will indicate better Vo2, METs and aerobic and physical capacity in the participant.
Changes in the Dyspnoea after 36 training sessions | After 3 month of training (36 training sessions)
  Dyspnea is a respiratory difficulty that usually translates into shortness of breath. Dyspnea can be determined using the original Borg scale (Score from 0 to 20) or modified (Score from 0 to 10), in which the higher the number indicated by the participant, the higher the degree of dyspnea.

IPD SHARING:
Plan to Share IPD: No
Initially, it is an issue that depends on the hospital institution where the research was conducted due to the personal data of the patients and the confidentiality of the institution. Therefore, initially it would be to talk with the patients, the institution and all the researchers. Mainly with the clinic because it is a bit jealous with your information.